CLINICAL TRIAL: NCT01864772
Title: Phase II Multicenter Trial Evaluating First Line Carboplatin, 5-Fluorouracil and Cetuximab in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Cancer, Aged 70 and Over, Ranked as Fit (no Frailty) by Geriatric Assessment
Brief Title: Phase II Trial of Carboplatin, 5-FU and Cetuximab in Elderly Fit (no Frailty) Patients With Recurrent/Metastatic HNSCC
Acronym: ELANFIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC ELAN-FIT
Record Dates: First submitted 2013-05-21; First posted 2013-05-30 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Metastatic or Recurrent Head and Neck Squamous Cell Cancer
Keywords: HNSCC; Metastatic; Recurrent; Elderly; Geriatry
MeSH Terms: conditions — Neoplasm Metastasis; Squamous Cell Carcinoma of Head and Neck; Recurrence | interventions — Fluorouracil; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carbo, 5FU, Cetuximab (Experimental): 6 cycles (1 cycle = 21 days) of: carboplatin AUC 5, 5FU D1-4 1000mg/m²/d, every 21 days cetuximab weekly (400 mg/m² the first week of treatment and then 250 mg/m²/w)
  Maintenance by cetuximab 500 mg/m² every 2 weeks until progression or toxicity
  Interventions: Drug: Carbo, 5FU, Cetuximab

INTERVENTIONS:
Drug: Carbo, 5FU, Cetuximab — 6 cycles (1 cycle = 21 days) of: carboplatin AUC 5, 5FU D1-4 1000mg/m²/d, every 21 days cetuximab weekly (400 mg/m² the first week of treatment and then 250 mg/m²/w)
  Maintenance by cetuximab 500 mg/m² every 2 weeks until progression or toxicity

SUMMARY:
The aim of the trial is to evaluate the clinical benefit (efficacy, safety, preservation of autonomy) of cetuximab-carboplatin-5FU combination as first line treatment of recurrent or metastatic head and neck squamous cell carcinoma in patients over 70 years without frailty (after geriatric assessment).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 70 years
* patient enrolled in ELAN-ONVOCAL study and evaluated as fit (harmonious aging) by GERICO screening method for geriatric frailty
* life expectancy superior to 12 weeks
* creatinin clearance > ou equal to 50ml/mn calculated using Modification of Diet in Renal Disease (MDRD) formula
* hematologic function : absolute neutrophil count > 1.5 x 10^9/l, platelets > 100 x 10^9/l, hemoglobin > 9,5 g/dl
* liver function : total bilirubin inferior to 1,25 x Upper limit of normal (ULN), SGOT/SGPT inferior to 5 x ULN, PAL inferior to 5 x ULN
* PS < 2

The disease:

* histologically proven head and neck squamous cell carcinomas
* recurrent or metastatic. Visceral metastases or locoregional recurrence unsuitable for curative locoregional treatment: unsuitable for primitive tumor surgery due to local extension (evidently authorized for lymph nodes) and unsuitable for radiotherapy for primitive tumor (or already performed) due to metastatic dissemination and the absence of indication for re-irradiation of primitive tumor.
* Presence of at least one measurable lesion (defined by RECIST criteria) by CT scan or IRM
* asymptomatic cerebral metastases authorized

General:

* signed Informed Consent Form
* affiliated to the French social security system (or a beneficiary of this system) according to the provisions of the law of 9 August 2004

Exclusion Criteria:

* Previous systemic chemotherapy, except for chemotherapy as part of multimodal treatment for locally advanced cancer completed more than 6 months prior to study enrollment
* Known contraindication specific to one of study treatments (particularly cardiac for 5FU)
* Known dihydropyrimidine dehydrogenase deficiency (DPD deficiency).
* Patients considered as "unfit " (fragile) by GERICO screening method for geriatric frailty
* Irradiation within 4 weeks prior to study enrollment.
* Nasopharyngeal, rhinopharyngeal or maxillary sinus carcinoma.
* Presence of infection (infection requiring intravenous antibiotics), including tuberculosis and HIV infection (human immunodeficiency virus).
* Concomitant treatment with other antitumor immunotherapy or hormonal therapy.
* Other antitumor concomitant therapies.
* Prior treatment with EGFR-targeted therapy (epidermal growth factor receptor).
* Treatment with one of study drugs within 30 days prior to study enrollment.
* Presence of documented symptomatic brain or leptomeningeal metastases
* Clinically significant coronaropathy or antecedent myocardial infarction within 12 months prior to study enrollment or high-risk uncontrolled arrhythmias or uncontrolled heart failure.
* Medically uncontrolled arterial hypertension
* Other prior or concomitant cancer, with exception for carcinoma in situ of the uterine cervix, or for cutaneous basal cell carcinoma within 5 years prior to study enrollment.
* Presence of medical or physiological factors susceptible to modify patient compliance with study protocol and follow-up or Informed Consent Form signing.
* Known allergy or hypersensibility to monoclonal antibodies (bevacizumab, cetuximab), or to other chemotherapies of the study or to their excipients

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Objective response and acute toxicity | 1 month after the end of chemotherapy
  Objective tumor response at 12 weeks, safety (no grade 3, 4, 5 toxicities) and preservation of geriatric autonomy (absence of 2 or more points decrease on the Activities of Daily Living (ADL) scale) 1 month after the end of chemotherapy

SECONDARY OUTCOMES:
Best objective tumor response | 6 weeks after the end of treatment
  Best objective tumor response during treatment
Overall survival | 1 year after the end of treatment
  Overall survival
progression free survival | 1 year after the end of treatment
  progression free survival
Duration of response under cetuximab maintenance therapy | 1 year after the end of maintenance
  Duration of response under cetuximab maintenance therapy
Toxicity of cetuximab maintenance therapy | 3 months after the end of maintenance
  Toxicity of cetuximab maintenance therapy
autonomy | 1 month after the end of treatment
  Autonomy assessed by ADL and IADL scales during treatment and until 1 month after the end of treatment
Health related quality of life | 1 month after the end of chemotherapy
  Quality of life assessed by EORTC QLQ-C30 and QLQ-HN35 questionnaires

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital de la Dracénie, Draguignan
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Guigay J, Le Caer H, Ferrand FR, Geoffrois L, Saada-Bouzid E, Fayette J, Sire C, Cupissol D, Blot E, Guillet P, Pavillet J, Bozec L, Capitain O, Rolland F, Debourdeau P, Pointreau Y, Falandry C, Lopez S, Coutte A, Chatellier T, Dalloz P, Ortholan C, Michel C, Lacas B, Cheurfa N, Schwob D, Bourhis J, Mertens C, Auperin A; ELAN Group including Gustave Roussy, Unicancer GERICO and H&N groups, and GORTEC. Adapted EXTREME regimen in the first-line treatment of fit, older patients with recurrent or metastatic head and neck squamous cell carcinoma (ELAN-FIT): a multicentre, single-arm, phase 2 trial. Lancet Healthy Longev. 2024 Jun;5(6):e392-e405. doi: 10.1016/S2666-7568(24)00048-5. Epub 2024 May 14. PMID 38759667
- See also: GORTEC — http://www.gortec.fr/